CLINICAL TRIAL: NCT04744753
Title: Assisted Oocyte Activation (AOA) in Recurrent Fertilization Failure
Brief Title: AOA in Recurrent Fertilization Failure
Acronym: AOA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: MOHAMED BEHERY (Other)
Responsible Party: Sponsor-Investigator, MOHAMED BEHERY, Behery MA, Al-Azhar University
Organization: Al-Azhar University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202010454
Record Dates: First submitted 2021-02-04; First posted 2021-02-09 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Infertility Primary

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- study group (Active Comparator): . This group involved 75 patients with history of fertilization failure in which oocytes were activated by calcium ionophores
  Interventions: Drug: Calcium Ionophore A23187
- control group (No Intervention): This group involved 75 patients with history of fertilization failure in which oocytes were not activated by calcium ionophores

INTERVENTIONS:
Drug: Calcium Ionophore A23187 — Calcium Ionophore A23187 is used in laboratories to increase intracellular Ca2+ levels in intact cells. It also uncouples oxidative phosphorylation, the process cells use to synthesize Adenosine triphosphate which they use for energy. In addition, A23187 inhibits mitochondrial ATPase activity. A23187 also induces apoptosis in some cells (e.g. mouse lymphoma cell line, or S49, and Jurkat cells) and prevents it in others (e.g. cells dependent on interleukin 3 that have had the factor withdrawn).
  In IVF field, Ca Ionophore can be used in case of low fertilization rate after ICSI procedure, particularly with Globozoospermia (Round Head sperm syndrome), Ca Ionophore will replace absence of sperm acrosom, and plays role in oocyte activation after ICSI. Recommended use is 0.5 microgram/ml twice for 10 min interrupted with fresh media with 30 min incubation, followed with regular injected eggs culture for IVF.
  Other Names: non
  Arms: study group

SUMMARY:
Background: Despite the high success rate of ICSI, total fertilization failure still occurs in 1-3% of all ICSI cycles and can recur in subsequent cycles, even when a sufficient number of oocytes and motile spermatozoa are available. Several reports show that the majority of couples suffering from ICSI failure benefit from the application of ICSI combined with assisted oocyte activation. A variety of artificial activating methods is used in human assisted reproduction treatment, including physical, mechanical or chemical stimuli, which provoke one or more calcium rises in the oocyte cytoplasm. Study Design: Randomized controlled trial. Setting: A university fertility center. Methods: 150 infertile patients who underwent ICSI and all had history of recurrent fertilization failure. The patients were randomly allocated into 2 equal groups. Group1=75 patients who underwent ICSI without oocyte activation. Group2 patients =75 and underwent ICSI Patient underwent ICSI with oocyte activation. Reproductive outcomes were compared between both groups. Results: there were significant differences between groups regarding number of oocytes retrieved, number of mature oocyte, fertilization rate and pregnancy rate. Conclusion: Assisted oocyte activation with calcium ionophore results in significant improvement in the fertilization, cleavage and pregnancy rates after ICSI.

DETAILED DESCRIPTION:
This study is a randomized controlled trial included 150 ICSI patients with history of recurrent fertilization failure. Patients had undergone ICSI trials in ART unit, Al-Azhar University, Cairo, Egypt, from July 2017 to November 2018. The study was approved by the university medical ethical committee (under registry number 202010454) and all couples had signed a written consent before initiation of the study and the treatment cycles. AOA candidate couples were counseled regarding the procedure. The patients were selected according to the following criteria:

Inclusion Criteria: -

1. Age between 20 and 40 years old.
2. Cases with history of total fertilization failure in previous ICSI cycles
3. Oocytes with normal morphology.
4. Male factor infertility. Exclusion Criteria: - Abnormal oocyte morphology degenerated or immature oocytes.

Two groups were randomly designated:

The first Group: The oocytes were treated by calcium ionophore. This group involved 75 ICSI cycles.

The Second Group: Oocytes were not treated by calcium ionophore. This group involved 75 ICSI cycles.

Methods:

1. Ovarian stimulation:

   All women received ovarian stimulating drugs according to the ART protocols (long agonist, flare up or antagonist protocols). Deca 0.1 was given s.c. daily, for down-regulation in short and long protocol while cetrotide 0.25 was given s.c. daily for down-regulation in antagonist protocol. Follicular development was monitored by ultrasound scanning and serum estradiol. Patients received 10,000 IU of Human Chronic Gonadotrophin (HCG) when most of the follicles measured more than 17-20 mm in diameter.
2. Semen preparation:

   • The husband was asked to submit a semen sample in a sterile plastic container after a 2 to 3-day period of abstinence and about 2 hours before the ICSI procedure. The specimen container must be clean, sterile and wide mouthed to minimize collection error.
3. Oocyte retrieval:

   * Under general anesthesia, the oocytes were aspirated by a specialized, ultrasound-guided needle (Labotect aspiration catheter, Germany) at 34-36 h after HCG injection. Warmed HEPES buffered medium (Irvine Scientific, Irvine, CA, USA) was used for handling and washing of oocytes.
   * After ICSI, the whole injected oocytes were washed with Global total Fertilization Medium (Global pharm, Life Global, Brussels, Belgium, Europe) and the patients were randomly allocated into two equal groups (75 patients each) by using computer-based randomization program. Group one in which, the injected oocytes were transferred to a medium that contain 10 µmol of calcium ionophore (GM508 Cult-Active, Gynemed, Germany) and were incubated for 10 minutes, then again oocytes were washed with Global total Fertilization Medium (Global pharm, Life Global, Brussels, Belgium, Europe) and were incubated at 37°C in 6% CO2. In group two, the injected oocytes were not submitted to calcium ionophore activation.
   * 18 hours after injection, the whole injected oocytes in both groups were evaluated for fertilization, cleavage and quality at the day of embryo transfer (ET).

Embryo Transfer

• After ET, luteal phase support was conducted (intramuscularly progesterone injection 100 mg daily) for 14 days until pregnancy test.

After data collection, both groups were compared regarding oocyte number, oocyte fertilization rate, number and quality of embryos, implantation rate and clinical pregnancy rate.

ELIGIBILITY:
Inclusion Criteria:

* (1) Age between 20 and 40 years old. (2) Cases with history of total fertilization failure in previous ICSI cycles (3) Oocytes with normal morphology.

Exclusion Criteria:

* (1) Abnormal oocyte morphology degenerated or immature oocytes. (2) Husbands with spermatogenic arrest or Sertoli/Leydig cells only.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2017-07-15 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2018-11-17 (Actual)

PRIMARY OUTCOMES:
fertilization rate | one and half year for all patients
  the number of reproduced embryos divided by the number of fertilized oocytes

SECONDARY OUTCOMES:
Pregnancy rate | one and half year for all patients
  the number of clinically pregnant women divided by the number of total patients undergoing ICSI procedures in the same group

CONTACTS AND LOCATIONS:
Overall Officials: doaa DA aswad, Master, Principal Investigator — specialist of obstetrics and gynecology
Locations (1):
- Al-Azhar University, Cairo, Nasr City, Egypt

IPD SHARING:
Plan to Share IPD: No